CLINICAL TRIAL: NCT05532930
Title: An Exploratory Study of Using Magnetic Resonance Prognostic Imaging Markers for Radiotherapy In Patients With Cervix Cancer
Brief Title: An Exploratory Study of Using Magnetic Resonance Prognostic Imaging Markers for Radiotherapy In Patients With Cervix Cancer (EMPIRIC Study)
Acronym: EMPIRIC
Status: Recruiting | Type: Observational
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Collaborators: University of Manchester (Other); Brunel University (Other)
Responsible Party: Sponsor
Other Study IDs: RD2021-29
Record Dates: First submitted 2022-09-05; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumour tissue samples at diagnosis and point of brachytherapy Peripheral blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with cervical cancer that has not spread to other parts of the body can be cured with radiotherapy. One of the reasons radiotherapy can fail is because there are areas within the tumour that have a poor oxygen supply which makes them resistant to radiotherapy. This study aims to assess if it is feasible using special types of magnetic resonance imaging (MRI) - multi-parametric (MP) MRI to identify areas of low oxygen within the tumour so a higher dose of radiation can be given specifically to these areas to overcome the resistance and potentially improve cure rates without increasing side effects.

DETAILED DESCRIPTION:
The study is an early exploratory study which will use MP MRI to predict which patients with locally advanced cervical cancer are likely to respond less well to chemoradiotherapy treatment, identify those patients and then intervene.

Hypoxia (deprivation of oxygen supply at tissue level) has long been shown to be a major cause of radiation resistance in various tumour sites and has been shown to be a harmful factor in cervical cancer and is associated with poor outcomes for patients. The aim of the study is to scan patients using different MP MRI sequences, each of which will measure different things, including blood flow, tumour necrosis and oxygen levels to determine hypoxia. This will be the first study to use the 3 different types of MRI scan (Diffusion Weighted - DWI, Dynamic Contrast Enhanced - DCE and Blood Oxygen Level Dependent - BOLD) at 3 different time points during the whole course of chemoradiotherapy.

The first scans will be prior to chemoradiotherapy treatment, the second set will be in week 2 and the final set in week 5. The imaging parameters from the MP MRI scans will be used as a surrogate markers of hypoxia. If high levels of hypoxia is identified using MP MRI, a prognostic imaging biomarker model can be developed to predict treatment outcomes of patients with locally advanced cervical cancer after chemoradiotherapy.

This study has potential to benefit all patients with locally advanced cervical cancer undergoing radical radiotherapy through the provision of more robust risk stratification. Improved risk stratification will result in more personalised treatment of better quality leading potentially to more cures and less side effects. As reported by Cancer Research UK, 3200 women are diagnosed with cervical cancer each year in the UK. 40% of these women are treated with radical radiotherapy, all of whom may benefit from the outputs of this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed FIGO stage Ib2-IVa squamous, adeno or adenosquamous carcinoma of the cervix.
* Clinically and/or radiographically documented measurable disease with at least one site of disease unidimensionally measurable as per RECIST 1.1
* All detectable disease including pelvic/para-aortic nodes encompassable within radical high-dose radiation field
* Deemed suitable and fit for radical chemoradiation
* ECOG performance status 0 - 1
* Aged 18 and over
* Documented negative pregnancy test (if applicable)
* Capable of providing written or witnessed informed consent according to ICH/GCP and national/local guidelines prior to registration

Exclusion Criteria:

* Previous pelvic malignancy (regardless of interval since diagnosis)
* Previous malignancy not affecting the pelvis (except basal cell carcinoma of the skin) where disease free interval is less than 10 years
* Evidence of distant metastasis i.e. any non-nodal metastasis beyond the pelvis
* Previous pelvic radiotherapy
* Prior diagnosis of Crohn's disease or Ulcerative colitis
* Uncontrolled cardiac disease (defined as cardiac function which would preclude hydration during cisplatin administration)
* Previous record of allergic reaction to Gadolinium-based contrast media and any other contra-indication to magnetic resonance imaging (MRI)
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the study
* Participation in any interventional trials

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Female participants
Study Population: Participants with locally advanced cervical cancer
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-08-05 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
To determine if multi-parametric MRI (MP MRI) can be used to predict progression-free survival of patients with locally advanced cervical cancer after chemoradiotherapy. | 1 and 2 years
  Progression-free survival measured by number of patients with local, distant and nodal progression
To determine if multi-parametric MRI (MP MRI) can be used to predict overall survival of patients with locally advanced cervical cancer after chemoradiotherapy. | 1 and 2 years
  Overall survival measured by number of patients with overall survival

SECONDARY OUTCOMES:
Temporal changes in MP MR parameters during chemoradiotherapy and the identification of a prognostic imaging biomarkers. | 2 years
  Parameters measured: Extravascular extracellular space volume fraction Ve (%), Transfer constant Ktrans (min-1), Rate Constant kep (min-1), Blood volume fraction vp (%), Apparent diffusion coefficient ADC (um2/sec), BOLD-based reversible transverse relaxation rate R2* (sec-1), Relaxation times (sec-1), 2nd order Haralick textural radiomic features

OTHER OUTCOMES:
Molecular markers correlated with imaging parameters and evaluated independently and in combination with respect to prognostic impact. | 2 years
  Tissue samples will assess immunohistochemical markers of hypoxia:
  (CA IX, GLUT-1), vascularity (VEGF) and epithelial mesenchymal transition(CD44, SOX-2).
  Blood samples - Circulation Tumour Cells (CTCs) will be classified into three subpopulations with respect to metastatic potential using epithelial mesenchymal transition markers: epithelial CTCs (EpCAM or CK8), mesenchymal CTCs (vimentin or TWIST) and mixed phenotype CTCs (both markers). The CTC phenotype ratio at various timepoints will be correlated with imaging parameters and evaluated independently and in combination with respect to prognostic impact.

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Vernon Cancer Centre, Northwood, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdul-Latif M, Chowdhury A, Tharmalingam H, Taylor NJ, Lakhani A, Padhani A, Hoskin P, Tsang Y. Exploratory study of using Magnetic resonance Prognostic Imaging markers for Radiotherapy In Cervix cancer (EMPIRIC): a prospective cohort study protocol. BMJ Open. 2024 Apr 18;14(4):e077390. doi: 10.1136/bmjopen-2023-077390. PMID 38637128